CLINICAL TRIAL: NCT02188199
Title: Clinical Care Continuum (C3) Total Joint Patient Registry
Brief Title: C3 Total Joint Patient Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DC2 Healthcare (Industry)
Collaborators: Clinical Care Continuum (C3) Foundation (Unknown); National Research Independent Operations Management (Other)
Responsible Party: Sponsor
Other Study IDs: C3 1001
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Knee Replacement; Hip Replacement
Keywords: Hip; Knee; Hip replacement; Knee replacement; Total Joint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Knee Replacement: Patients undergoing knee replacement surgery
- Hip Replacement: Patients undergoing hip replacement

SUMMARY:
This study will assess the efficacy of products, implants, and procedures for knee and hip replacement.

DETAILED DESCRIPTION:
This registry will prospectively collect a core set of data on patients undergoing knee or hip replacement. This registry will include a variety of different products, implants, technologies and procedures. The registry will also collect any adverse events/complications that occur during or following these surgeries. This database can also be utilized in the future to answer research questions, by retrospectively going back through the data. This information also may go to insurance companies or hospitals for quality measurement and metrics reporting. The data will be utilized to develop strategic treatment pathways that will improve patient care. Ultimately, the goal of the registry is to enhance the understanding of treatment associated with knee and hip replacement and the resulting patient outcomes. The registry will also be used to provide quality measurement and metrics reporting.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Undergoing knee or hip replacement
* Subject is likely to follow standard of care post-operative follow up for at least 1 year

Exclusion Criteria:

* Inability to complete follow-up visits or required questionnaires
* Inability to provide informed consent without a legally authorized representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will come from cohorts of patients undergoing either knee or hip replacement in accordance with a nationwide multicenter observational study design. Eligibility criteria require only that patients are undergoing knee or hip replacement, are able to sign informed consent and are 18 years of age or older. Approximately 10,000 patients will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in Hip disability and Osteoarthritis Outcome Score (HOOS) from baseline at 3 months | baseline and 3 months
  Assessment of hip symptoms and disability to be taken at baseline and 3 months after surgery
Change in Hip disability and Osteoarthritis Outcome Score (HOOS) from baseline at 6 months | baseline and 6 months
  Assessment of hip symptoms and disability to be taken at baseline and 6 months after surgery
Change in Hip disability and Osteoarthritis Outcome Score (HOOS) from baseline at 1 year | baseline and 1 year
  Assessment of hip symptoms and disability to be taken at baseline and 1 year after surgery
Change in Knee injury and Osteoarthritis Outcome Score (KOOS) from baseline at 3 months | baseline and 3 months
  Assessment of knee symptoms and disability to be taken at baseline and 3 months after surgery
Change in Knee injury and Osteoarthritis Outcome Score (KOOS) from baseline at 1 year | baseline and 1 year
  Assessment of knee symptoms and disability to be taken at baseline and 1 year after surgery
Change in Knee injury and Osteoarthritis Outcome Score (KOOS) from baseline at 6 months | baseline and 6 months
  Assessment of knee symptoms and disability to be taken at baseline and 6 months after surgery

SECONDARY OUTCOMES:
Adverse Events at time of surgery | Time of surgery
Adverse Events at 6 weeks after surgery | 6 weeks after surgery
  within 6 weeks but not less than 1 week after surgery
Adverse Events at 3 months after surgery | 3 months after surgery
Adverse Events at 6 months after surgery | 6 months after surgery
Adverse Events at 1 year after surgery | 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- DC2 Healthcare, Nashville, Tennessee, United States

REFERENCES:
- See also: DC2 Healthcare — http://www.dc2healthcare.com
- See also: NRIOM — http://www.nriom.com/